CLINICAL TRIAL: NCT00404183
Title: A Randomized, Multi-center, Double-blind Study Comparing the Analgesic Efficacy and Safety of Extended Release Hydrocodone/Acetaminophen and Placebo in Subjects With Osteoarthritis
Brief Title: A Study Comparing the Analgesic Efficacy and Safety of Extended Release Hydrocodone/Acetaminophen (Vicodin® CR)and Placebo in Subjects With Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Victor Jorden, MD, Abbott
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M03-643
Record Dates: First submitted 2006-11-26; First posted 2006-11-28 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Pain
Keywords: Pain associated with osteoarthritis
MeSH Terms: conditions — Pain | interventions — Acetaminophen; Hydrocodone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- hydrocodone/acetaminophen extended release (Experimental)
  Interventions: Drug: Extended-Release Hydrocodone/Acetaminophen
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Extended-Release Hydrocodone/Acetaminophen — 2 tablets BID
  Other Names: ABT-712; hydrocodone/acetaminophen extended release
  Arms: hydrocodone/acetaminophen extended release
Drug: Placebo — 2 tablets BID
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness (level of pain control) and safety of the administration of Extended Release Hydrocodone/Acetaminophen with placebo over a 5-week dosing period in patients with osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ages 21 to 75
* Has osteoarthritis of the hip or knee
* Requires therapeutic doses of medications for osteoarthritis
* If female, must be of non-childbearing potential or practicing birth control
* Has sufficient pain to justify the use of round-the-clock opioids

Exclusion Criteria:

* Has received certain types of procedures or received certain medications for osteoarthritis within a specific timeframe
* Has certain medical conditions which may interfere with pain assessments
* Is allergic to or has a serious reaction to hydrocodone, other opioids, or acetaminophen
* Has had certain infections, injuries or illnesses within the last month
* Has had major abdominal surgery, certain diseases that may cause intestinal narrowing, or has a history of constipation, diarrhea or nausea and vomiting
* Is receiving chemotherapy, or has been diagnosed with certain cancers within the past 5 years
* Has a history of major psychiatric disorders or requires treatment with certain drugs for depression
* Cannot discontinue pain medications, even for a short time, prior to the study start

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2004-08; Primary Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Pain intensity difference from baseline to final assessment using the VAS scale (100 mm, 0 being "no pain" and 100 being "worst pain imaginable"). | 4 weeks
  Arthritis Pain Intensity measured by a 100mm Visial Analog Scase (VAS)

SECONDARY OUTCOMES:
WOMAC Osteoarthritis Index, SF36 | 4 weeks
  Osteoarthritis Index

CONTACTS AND LOCATIONS:
Overall Officials: Rita Jain, MD, Study Director — Abbott